CLINICAL TRIAL: NCT04100668
Title: Evaluation of Sensifree's Alpha Sensor Signal Morphology in Comparison to Invasive Radial Arterial Line Pressure Waveform and PPG Signal Morphology
Brief Title: Evaluation of Sensifree's Alpha Sensor Signal Morphology Compared to Arterial Line and PPG Signal Morphologies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sensifree Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PR2017-240
Record Dates: First submitted 2018-03-28; First posted 2019-09-24 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Blood Pressure Measurement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Data collection (Experimental): Comparing radial arterial line, Sensifree's Alpha sensor and PPG sensor pressure waveforms
  Interventions: Device: Sensifree's Alpha sensor; Device: Arrow® arterial catheterization kit (Teleflex); Device: GE Datex-Ohmeda Oxy-F Finger Clip Pulse Oximeter Sensor

INTERVENTIONS:
Device: Sensifree's Alpha sensor — RF based, wrist mounted sensor, that acquires a high fidelity signal originating at the radial artery, and constructs a pressure waveform
Device: Arrow® arterial catheterization kit (Teleflex) — Invasive monitoring of blood pressure via catheterization of the radial artery, displaying a continuous pressure waveform
Device: GE Datex-Ohmeda Oxy-F Finger Clip Pulse Oximeter Sensor — PPG based, fingertip mounted sensor, that measures the oxygen level (oxygen saturation) of the blood and generates a waveform

SUMMARY:
The purpose of the protocol is to compare Sensifree Alpha sensor signal morphology, measured at the radial artery, to an invasive arterial line pressure signal and the oxygen saturation as read by a pulse oximeter.

The study will be split into two phases: the first phase will collect data for morphology analysis and algorithm development, the second phase will compare device performance to the reference invasive blood pressures. A secondary objective is to evaluate signal morphology changes due to changes in subject arm position.

DETAILED DESCRIPTION:
This study is a single-center, non-randomized study with a maximum of 50 subjects. The duration of the study for each subject test is expected to take approximately 3 hours: 1 hour for screening (Visit 1) and 2 hours for data collection (Visit 2).

Data Collection, Visit 2, will be divided into two phases. Phase 1 will use up to 20 subjects with the goal of collecting data for algorithm and sensor development. No requirements for certain blood pressure populations are required for Phase 1. Once the analysis of the Phase 1 results is complete, Phase 2 will use up to 30 subjects with the following requirements to test multiple blood pressure populations:

* No more than 25% will be normotensive
* At least 60% of the subjects will be hypertensive
* At least 15% of the subjects will be hypotensive

Visit 1- Screening Screening will be identical for both phases of the study. Subjects will be screened for per the inclusion criteria, assuring the subject will be a good candidate for the data collection portion of the study. If the subject does not meet the inclusion criteria they will not be invited to participate in Visit 2. During screening, the subject's wrist circumference will be recorded and measured for each arm. The clinician will perform auscultatory blood pressure measurements on both arms to determine the lateral systolic and diastolic blood pressure difference per Procedure 5.2.4.3.1. in the International Standards Organization (ISO) 81060-2:2013. Using ultrasound, the clinician will also determine if the subject has any bifurcations in the radial artery of each arm. Finally, the investigation devices will be place on both wrists of the subject to determine if adequate signal can be detected. If the subject meets all the inclusion criteria for screening they will be invited to participate in the data collection portion of the study during Visit 2.

Visit 2- Screening Visit 2, the data collection portion of the study, will begin with the volunteer test subject lying in the supine position. The subject will be reminded they may withdraw from the study at any time. The subject will have the investigational device, ECG sensors, and a pulse oximetry sensor placed on them for data collection and to monitor their safety for the duration of the study. An arterial line will be placed in the radial artery, contralateral to the investigational device, under sterile conditions by a physician. To begin data collection; 10 minute periods of simultaneous invasive data from the arterial line and the non-invasive signal from the investigational device will be recorded. Once the supine recording sessions are complete, the subject will be raised to a seated position and the pressure transducer will be recalibrated. The subject will then vary both their arm positions simultaneously from heart level, to above heart level, and to below heart level to record the changes in pressure due to movement.

Once all data has been collected, the radial arterial catheter will be removed by the physician and constant pressure held on the arterial puncture for a minimum of 10 minutes. The clinician will review any final questions with the subject, the subject will be provided with phone numbers for questions pertaining to the participation in this study or research-related injury or reaction post study. Follow-up with each subject will be conducted within 5 days following participation in the study and will be conducted via telephone, text, or email.

ELIGIBILITY:
Inclusion Criteria:

* General:

  * Subject must have the ability to understand and provide written informed consent
  * Subject must be willing and able to comply with study procedures and duration
* Screening and Phase 1:

  * Subject is from 20 to 55 years old.
  * Subject has wrist circumference size within 145 and 220mm for both arms.
  * Subjects with lateral blood pressure difference (auscultatory cuff based measurement) is less than: 15 mmHg for systolic blood pressure. 10 mmHg for diastolic blood pressure.
  * Subjects with investigational device signal quality higher than a predefined value
  * Subjects with similar investigational devices signals between their two arms.
* Phase 2 (all requirements as Phase 1 except):

  * Subject is from 20 to 85 years old.
  * At least 60% of subjects will have hypertensive blood pressure values (goal) (systolic >140 mmHg and/or diastolic >90 mmHg)
  * At least 15% of subjects will have hypotensive blood pressure values (goal) (systolic <110 mmHg and/or diastolic <60 mmHg).
  * No more than 25% of subjects will have normotensive blood pressure values (goal) (systolic from 110 to 140 mmHg and/or diastolic from 60 to 90 mmHg).

Exclusion Criteria:

* Subject with a BMI over 39
* Deformities or abnormalities that may prevent proper application of the device under test
* Females who are pregnant, who are trying to get pregnant, or have a urine test positive for pregnancy on the day of the study
* Subjects with known respiratory conditions such as: (self-reported)

  * uncontrolled / severe asthma,
  * flu,
  * pneumonia / bronchitis,
  * shortness of breath / respiratory distress,
  * respiratory or lung surgery,
  * emphysema, COPD, lung disease
* Subjects with known heart or cardiovascular conditions such as: (self-reported, except for blood pressure and ECG review)

  * have had cardiovascular surgery
  * have cardiac pacemakers and/or automatic internal cardio-defibrillator
  * Chest pain (angina)
  * Abnormal pulse pressure
  * previous heart attack
  * blocked artery
  * unexplained shortness of breath
  * congestive heart failure (CHF)
  * history of stroke
  * transient ischemic attack
  * carotid artery disease
  * myocardial ischemia
  * myocardial infarction
  * cardiomyopathy
  * Subject with a heart rate of less than 45 BPM
* Self-reported health conditions as identified in the Health Assessment Form (self- reported)

  * diabetes,
  * uncontrolled thyroid disease,
  * kidney disease / chronic renal impairment,
  * history of seizures (except childhood febrile seizures),
  * epilepsy,
  * history of unexplained syncope,
  * recent history of frequent migraine headaches,
  * recent head injury
  * cancer / chemotherapy
* Subjects with known clotting disorders (self-reported)

  * history of bleeding disorders or personal history of prolonged bleeding from injury
  * history of blood clots
  * hemophilia
  * current use of blood thinner: prescription or daily use of aspirin
* Subjects with severe contact allergies to standard adhesives, latex or other materials found in pulse oximetry sensors, ECG electrodes, respiration monitor electrodes or other medical sensors (self-reported)
* Subjects with a contact allergy to ultrasound gel.
* Subjects with prior or known allergies to iodine or lidocaine (or similar pharmacological agents, e.g. Novocaine)
* Failure of the Perfusion Index Ulnar/Ulnar+Radial Ratio test
* Subject is intoxicated during the time of the visit, or was intoxicated within 24 hours prior to study visit, as reported by the subject, or per study staff judgment.
* Other known health condition, should be considered upon disclosure in health assessment form
* Subjects with heart rate below 45 BPM.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2017-09-26 (Actual); Primary Completion 2017-09-29 (Actual); Study Completion 2017-09-29 (Actual)

PRIMARY OUTCOMES:
Comparison of signals acquired from the investigational device, pulse oximeter, and arterial line | Three hours
  BP waveform will be acquired form three sources (PPG, A-line and investigational device),data will be statistically analyzed to find the correlations between the different sources of BP waveform

SECONDARY OUTCOMES:
Evaluation of waveform signal changes with different arm positions | Three hours
  Recordings will be made using the investigational device with different position of the subject arm to assess the effect of the arm positions (arm up, down and in chest level) over the acquired BP waveform signal

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Ruiz Cabrera, M.D, Principal Investigator
Locations (1):
- Clinimark Lab, Louisville, Colorado, United States

IPD SHARING:
Plan to Share IPD: No